CLINICAL TRIAL: NCT04272060
Title: Ultra-High Resolution CT vs. Conventional Angiography for Detecting Hemodynamically Significant Coronary Artery Disease - The Core-PRECISION MULTI-CENTER STUDY
Brief Title: Ultra-high-resolution CT vs. Conventional Angiography for Detecting Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00209321
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary heart disease; coronary angiography; CT angiography; cardiac catheterization
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — Computed Tomography Angiography

STUDY DESIGN:
Intervention Model Description: All patients are being asked to undergo a research CT scan in addition to the clinically prescribed invasive coronary angiogram (each patient is the patient's own "control" for the diagnostic test)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CT Angiography (Experimental): Research CT angiography.
  Interventions: Diagnostic Test: CT angiography
- Conventional Angiography (Active Comparator): Standard medical care which includes cardiac catheterization and invasive coronary angiography.
  Interventions: Diagnostic Test: Invasive coronary angiography

INTERVENTIONS:
Diagnostic Test: CT angiography — Diagnostic CT angiography
  Arms: CT Angiography
Diagnostic Test: Invasive coronary angiography — Diagnostic invasive coronary angiography
  Arms: Conventional Angiography

SUMMARY:
Cardiac catheterization with invasive coronary angiography is the gold standard for determining the presence or absence of significant coronary heart disease (CHD). However, cardiac catheterization is costly and, as an invasive procedure, it is associated with some risk of adverse events, rarely even stroke, myocardial infarction, or death. Recent advances in multi-detector computed tomography angiography (CTA) have allowed rapid, noninvasive coronary artery imaging in patients with suspected CHD. CTA generally yields high accuracy for identifying patients with CHD when compared to cardiac catheterization. However, diagnostic accuracy is reduced in the setting of severe coronary artery calcification and coronary stents due to its inferior spatial resolution compared to cardiac catheterization. Because high-risk patients often have severe coronary calcification or stents, the application of CTA has been particularly limited in this important patient group. Recently, an ultrahigh-resolution CT scanner was released which has shown promise to overcome the limitation of conventional CTA in the setting of severe coronary artery calcification or stents. This ultrahigh-resolution "precision" CT scanner (UHR-CT) contains detector rows with half the width than currently available systems (0.25 mm vs. 0.5 mm) resulting in approximately twice the spatial resolution.

The purpose of this investigation is to test the hypothesis that high-resolution CTA is not inferior to the current standard of cardiac catheterization for identifying significant CHD in patients with high-risk characteristics, including severe coronary artery calcification and coronary stents.

The investigators propose to enroll 50 patients over 24-30 months in this investigation as part of a multicenter study. Patients referred for cardiac catheterization with known CHD and suspected obstructive coronary artery stenosis will be included. All patients will undergo both cardiac catheterization and UHR-CT for determining significant CHD as defined by coronary functional assessment. The primary end point will be the diagnostic accuracy by area-under-curve (AUC) method for identifying patients with hemodynamically significant CHD.

DETAILED DESCRIPTION:
1. Objectives:Primary Objective The primary objective of this study is to generate preliminary data in support of the hypothesis that noninvasive UHR-CT is not inferior to invasive coronary angiography by cardiac catheterization for identifying patients with hemodynamically significant CHD.

Secondary Objectives Secondary objectives include testing the diagnostic accuracy of UHR-CT vs. cardiac catheterization on a vessel and segment-based analysis, comparison of UHR-CT Fractional Flow Reserve (FFR) to conventional angiography, and comparison of adverse events and radiation doses between the CT and conventional angiography groups.

Patient-Based Hypotheses

1. Diagnostic accuracy of UHR-CT using visual assessment of coronary artery disease is non-inferior to invasive, conventional coronary angiography for identifying patients with hemodynamically significant CHD defined by an FFR or QFR-value of <0.8 in at least one vessel of 2.0 mm or larger in diameter.
2. Diagnostic accuracy of UHR-CT using quantitative assessment of coronary artery disease is non-inferior to invasive, conventional coronary angiography for identifying patients with hemodynamically significant CHD defined by an FFR-value of <0.8 in at least one vessel of 2.0 mm or larger in diameter.
3. UHR-CT coronary angiography is associated with lower radiation dose than conventional, invasive coronary angiography.
4. UHR-CT coronary angiography is associated with lower adverse effects than conventional, invasive coronary angiography.

Vessel Based Hypotheses

1. Diagnostic accuracy of UHR-CT using visual assessment of coronary artery disease is non-inferior to invasive, conventional coronary angiography for identifying vessels with hemodynamically significant CHD defined by an QFR-value of <0.8 in a vessel of 2.0 mm or larger in diameter.
2. Diagnostic accuracy of UHR-CT using quantitative assessment of coronary artery disease is non-inferior to invasive, conventional coronary angiography for identifying vessels with hemodynamically significant CHD defined by an FFR-value of <0.8 in a vessel of 2.0 mm or larger in diameter.

   Lesion-Based Hypotheses
3. Diagnostic accuracy of UHR-CT using visual assessment of coronary artery disease is non-inferior to invasive, conventional coronary angiography for identifying lesions with hemodynamically significant CHD defined by an QFR-value of <0.8 in a vessel of 2.0 mm or larger in diameter.
4. Diagnostic accuracy of UHR-CT using quantitative assessment of coronary artery disease is non-inferior to invasive, conventional coronary angiography for identifying lesions with hemodynamically significant CHD defined by an QFR-value of <0.8 in a vessel of 2.0 mm or larger in diameter.

2. Background: Cardiac catheterization with invasive coronary angiography has remained the gold standard for determining the presence or absence of significant coronary luminal stenosis despite its limited accuracy compared to the standard of intravascular ultrasound. Because of the inherent risks involved with this invasive procedure (e.g., stroke, myocardial infarction, death or need for emergency surgical intervention) with a major complication rate of 1-2%), and considerable costs, non-invasive assessment of coronary artery disease would be preferred. Advances in multi-detector computed tomography angiography (CTA) have made the non-invasive imaging of the coronary arterial lumen and wall feasible. Numerous studies have since demonstrated good accuracy of CTA to identify patients with obstructive coronary artery disease. However, studies also demonstrated that CTA's diagnostic accuracy is only modest in patients with severe coronary artery calcification or stents, representing a major limitation of the technology. This limitation is due to fair spatial resolution and associated image artifacts in the setting of an attenuation-based image reconstruction algorithm. In this situation, high density structures, such as calcium or metal, will disproportionally dominate information derived from an affected image voxel leading overrepresentation of these structures on image display (partial volume effect).

Recently, an ultrahigh-resolution CT scanner has been released which has shown promise to overcome the limitation of conventional CTA in the setting of severe coronary artery calcification or stents. This ultrahigh-resolution "precision" CT scanner (UHR-CT) contains detector rows with half the width than currently available systems (0.25 mm vs. 0.5 mm) resulting in approximately twice the spatial resolution. It is likely that this improvement will lead to improved diagnostic accuracy in high-risk patients. To conclusively test this hypothesis, a larger, multi-center study is required. The purpose of this investigation is to test the feasibility of such study and to generate initial data on the hypothesis that high-resolution CTA is not inferior to the current standard of cardiac catheterization for identifying significant CHD in patients with high-risk characteristics.

3. Study Procedures

a) Study design: The CORE-PRECISION MULTI-CENTER study is a prospective diagnostic accuracy study at three international sites comparing the diagnostic accuracy of UHR-CT to conventional, invasive coronary angiography by cardiac catheterization for the presence of hemodynamically significant CHD in 150 patients with high pretest probability of obstructive CHD. The enrollment at all centers is expected to commence in the summer of 2022: Johns Hopkins Hospital and Johns Hopkins Bayview Medical Center, Baltimore, USA, Iwate University Medical Center, Iwate, Japan, and Einstein Medical Center, Sao Paulo, Brazil. Sites will obtain approval from the local Institutional Review Board and all patients will sign informed consent prior to participation Each study site is expected to enroll 50 participants. Enrollment has been ongoing since November of 2019 at Johns Hopkins University as part of a pilot study using the same protocol with minor variations. For each participant, it is anticipated that the Screening Evaluation Periods will last less than 2 months and will be followed by the Imaging period (less than 60 days). All patients will be followed by additional 30 days after cardiac catheterization for occurrence of adverse events.

Screening-Evaluation Period: The screening period will begin when a patient is scheduled for a clinically indicated coronary angiogram. The protocol inclusion and exclusion criteria will be reviewed for each potential participant. Patients without history of Coronary Artery Disease (CAD) may enter an extended screening period that involves the first component of the CT imaging examination, namely the coronary calcium scan. If this scan shows a calcium score <400, these patients will be considered late screen failures, will not proceed to contrast-enhanced coronary CT angiography, and will be excluded from further participation in the trial. Patients with a calcium score of 400 or greater will proceed to coronary CT angiography and study participation.

If the patient appears to be eligible for the study based on the initial evaluation, informed consent will be obtained. Baseline information and medical history will be collected. Blood will be obtained at the time of CTA (during intravenous cannula [IV] placement) for laboratory testing of cholesterol profile and serum biomarkers. No genetic testing will be performed. The clinically indicated coronary angiogram will not be delayed to complete the research protocol. If the CTA scan cannot be scheduled prior to the clinically indicated coronary angiogram the patient will not be enrolled in the trial. Consented patients will continue to be evaluated for participation in the trial through the imaging period.

Imaging Period: The imaging period will consist of two tests: 1) ultra-high resolution CT (UHR-CT) angiography; 2) conventional coronary angiography (CTA). All enrolled patients referred for a clinically indicated catheterization will first a UHR-CT angiogram. All enrolled patients referred for a clinically indicated catheterization will first receive a UHR-CT angiogram to avoid conflict with coronary artery revascularization

UHR-CT Imaging: Patients will have one 18-20 gauge intravenous lines placed, preferably in an antecubital vein for contrast administration. The patient will be hydrated with normal saline intravenously (250 - 500 ml) prior to UHR-CT scanning. The patient will lie supine on the scanner table and be attached to a 12 lead electrocardiographic monitor and an automated blood pressure monitor. Baseline electrocardiogram (ECG), heart rate, and blood pressure will be recorded and reviewed by one of the study investigators. Due to resultant artifacts from precordial leads, the 12 ECG leads and electrodes will be removed and rhythm monitoring will continue using the 3-lead system attached to the scanners monitoring system during scanning. Patients may receive oral metoprolol and/or oral ivabradine 1-2 hours prior to the CT according to a hospital approved heart rate control algorithm. Specifically, if the heart rate (HR) is >70 beats per minute, 50 mg of oral metoprolol will be given along with 15 mg of oral ivabradine. If the heart rate is >65 but lower than 70 beats per minute, 25 mg of oral metoprolol will be given along with 15 mg of oral ivabradine. If the heart rate is >60 beats per minute but lower than 65 beats, only 15 mg of ivabradine is given. If HR remains >60 beats per minute after 60 minutes post initial dosing of metoprolol and ivabradine, a second doses of 25-50 mg oral metoprolol is given. Scout images for determining scanning range will be obtained in the anterior-posterior and lateral views. Patients with systolic blood pressure ≥100 will receive 0.4-1.2 mg sublingual nitroglycerin for vasodilation. The adequate calcium score scan protocol will be confirmed on the scanner for each participant prior to the initiation of the calcium score scan. Patients will then be asked to hold patients' breath (approximately 10-15 seconds) and non-contrast CT imaging will be performed starting just cranial to the coronary ostia and extending just caudal to the apex of the heart in order to obtain a coronary calcium score. To limit radiation exposure, a coronary calcium score will only be generated for patients who have not previously been stented as the presence of stents affects the accuracy of the calcium score. CT angiogram will then be performed to evaluate the coronaries using iodine contrast.

UHR-CT Protocol for Coronary Angiography

1. If no previous stents, coronary calcium scan will be performed using the following protocol:

   * No contrast.
   * CT Imaging: tube voltage = 120 kilovolt (kV), tube current = 150 milliAmpere (mA), gantry rotation speed = 0.230 seconds for half rotation, slice thickness = 0.25 mm, rows = 100, range = 144 mm. Estimated radiation dose = 0.5--2.0 milli-Sievert (mSv).
2. Coronary arterial imaging will be performed during a 4-6 ml/sec intravenous iodinated contrast infusion for a total volume of 60-120 ml. The automated bolus tracking feature will be used to judge contrast bolus arrival and optimize image quality.

Images will be prospectively triggered using ECG gating which reduces radiation exposure to the patient compared to retrospective gating. Tube voltage and current will be adjusted according to image noise characteristics during scout imaging. A tube setting of 120 kV with 580 mA will be required for most patients in the setting of severe calcification and/or stenting. Target exposure will be 70-80% of the R-R cycle for heart rate ≤60 bpm. Heart rate of 61-70 will require a widened exposure window of 65-85% of the R-R cycle. Gantry rotation will be 350 ms with a 160 x 0.25 mm collimation in super high resolution mode, requiring approximately 6.5 second scan time. The estimated range of radiation dose for CT coronary angiography will be 4.3.0-10.7 mSv depending on patient size and weight.

Total estimated radiation dose, including calcium scoring, bolus tracking, and CT coronary angiography, will therefore range between 4.8-12.7 mSv. For comparison, a standard nuclear stress test typically results in a radiation dose of 10-12 mSv to the patient. Diagnostic cardiac catheterization for conventional coronary angiography typically averages 12 mSv radiation dose.

A copy of the anonymized raw data (without any patient identifiers) will be forwarded to the CT Core Laboratory for analysis within 1 week of the scan. CT raw data and reconstructed data will be saved by the site for at least 5 years after completion of the study.

Within 3 weeks of the CTA, the CTA will be reviewed for non-cardiac findings by a locally qualified, institutionally approved radiologist, and reported. The investigator will report these findings to the patient's clinical physician and patient in a timely fashion preferably prior to or during the 30-day follow-up.

A pre-catheterization serum creatinine should be obtained post CTA (per local standard, or preferably > 2 days post CTA).

Conventional Coronary Angiography Patients will undergo patients' clinically indicated cardiac catheterization/coronary angiography, within 60 days of CT imaging with a recommended goal of completing all imaging within 30 days. A time window of ≥ 24-48 hours is recommended between CT imaging and conventional coronary angiography to minimize cumulative risk of contrast exposure from these two tests. Coronary angiography guidelines to obtain optimum angles and images for comparison will be enforced. Isocenter calibration will be performed for all studies to enable quantitative flow reserve (QFR) assessment. Intracoronary nitroglycerine will be administered (150-200 mcg) prior to first image of the left coronary artery system and right coronary artery. This is to standardize the vasomotor state of the coronary artery and eliminate any potential for catheter-induced changes (i.e., catheter induced spasm).

Fractional-flow-reserve (FFR) assessment may be performed as clinically indicated but not solely for research purposes. Coronary angiographic images will be saved in the universal DICOM format and forwarded to the Angiographic Core Laboratory for Quantitative Coronary Angiographic Analysis. Quantitative coronary analysis (QCA) will be performed using standard, validated analysis software from Medis Medical Systems (Medis QCA). QFR will be performed using a dedicated software (QFR, Medis Medical Imaging Systems).

A post-catheterization serum creatinine should be obtained per local standard, or preferably within 48-72h post invasive coronary angiogram.

Primary Objective The primary objective of this study is to generate preliminary data in support of the hypothesis that noninvasive UHR-CT is not inferior to invasive coronary angiography by cardiac catheterization for identifying patients with hemodynamically significant CHD.

Secondary Objectives Secondary objectives include testing the diagnostic accuracy of UHR-CT vs. cardiac catheterization on a vessel and segment based analysis, comparison of UHR-CT Fractional Flow Reserve (FFR) to conventional angiography, and comparison of adverse events and radiation doses between the CT and conventional angiography groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45-85 years with history of CHD will be asked to participate. History of CHD is defined as prior documentation of a coronary artery stenosis of 50% or greater by coronary angiography or by prior documentation of coronary artery revascularization by percutaneous coronary intervention (PCI). Women of child bearing potential must demonstrate a negative pregnancy test within 24 hours of the study CTA.
* Suspected obstructive coronary artery stenosis based on clinical history and/or noninvasive testing, prompting a clinical referral for invasive coronary angiography; and/or planned PCI within the next 60 days.
* Ability to understand and willingness to sign the Informed Consent Form.

Exclusion Criteria:

* Known allergy to iodinated contrast media
* History of multiple myeloma or previous organ transplantation
* Elevated serum creatinine (> 1.5mg/dl) or calculated creatinine clearance of < 60 ml/min (using the Cockcroft-Gault formula
* Atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third-degree heart block)
* Evidence of severe symptomatic heart failure (NYHA Class III or IV);
* Known or suspected moderate or severe aortic stenosis
* Previous coronary artery bypass or other cardiac surgery
* Patients without a history of CHD who had no or only mild coronary calcification on chest CT imaging within the past 5 years or had most recent coronary calcium scan with a score <400
* Suspected acute coronary syndrome
* Presence of any other history or condition that the investigator feels would be problematic

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with hemodynamically significant coronary heart disease | Up to 24 months
  The primary analysis will be a comparison of the diagnostic capability of the UHR-CT angiography to conventional coronary angiography at the patient level with the reference standard being coronary flow reserve assessment by either fractional flow reserve (FFR) or quantitative flow reserve (QFR). A positive patient will be defined as having at least one vessel with a flow reserve <0.8. If both assessments are available for the same vessel, the FFR will be used as reference.

SECONDARY OUTCOMES:
Number of coronary arteries with abnormal fractional flow reserve | Up to 24 months
  A positive vessel will be defined as having at least one stenosis with a flow reserve <0.8 (abnormal fractional flow reserve).
Radiation Dose | At the time of diagnostic procedure, up to 30 minutes
  Radiation dose (mSv) estimates for both CT and conventional angiography will be recorded and compared for both tests.
Number of adverse outcomes | Up to 24 months
  Adverse patient outcome defined as a composite outcome of death, stroke, myocardial infarction, acute renal failure, acute vascular injury, or major bleeding. This will be assessed separately for 24 hours after imaging and will be compared for CTA and conventional angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Armin A Zadeh, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data belong to sponsor who may or may not release data to other researchers

REFERENCES:
- [Result] Raff GL, Gallagher MJ, O'Neill WW, Goldstein JA. Diagnostic accuracy of noninvasive coronary angiography using 64-slice spiral computed tomography. J Am Coll Cardiol. 2005 Aug 2;46(3):552-7. doi: 10.1016/j.jacc.2005.05.056. PMID 16053973
- [Result] Arbab-Zadeh A, Miller JM, Rochitte CE, Dewey M, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic accuracy of computed tomography coronary angiography according to pre-test probability of coronary artery disease and severity of coronary arterial calcification. The CORE-64 (Coronary Artery Evaluation Using 64-Row Multidetector Computed Tomography Angiography) International Multicenter Study. J Am Coll Cardiol. 2012 Jan 24;59(4):379-87. doi: 10.1016/j.jacc.2011.06.079. PMID 22261160
- [Result] Wykrzykowska JJ, Arbab-Zadeh A, Godoy G, Miller JM, Lin S, Vavere A, Paul N, Niinuma H, Hoe J, Brinker J, Khosa F, Sarwar S, Lima J, Clouse ME. Assessment of in-stent restenosis using 64-MDCT: analysis of the CORE-64 Multicenter International Trial. AJR Am J Roentgenol. 2010 Jan;194(1):85-92. doi: 10.2214/AJR.09.2652. PMID 20028909
- [Result] Takagi H, Tanaka R, Nagata K, Ninomiya R, Arakita K, Schuijf JD, Yoshioka K. Diagnostic performance of coronary CT angiography with ultra-high-resolution CT: Comparison with invasive coronary angiography. Eur J Radiol. 2018 Apr;101:30-37. doi: 10.1016/j.ejrad.2018.01.030. Epub 2018 Feb 1. PMID 29571798
- [Result] Tanaka R, Yoshioka K, Takagi H, Schuijf JD, Arakita K. Novel developments in non-invasive imaging of peripheral arterial disease with CT: experience with state-of-the-art, ultra-high-resolution CT and subtraction imaging. Clin Radiol. 2019 Jan;74(1):51-58. doi: 10.1016/j.crad.2018.03.002. Epub 2018 Apr 5. PMID 29627067
- [Result] Einstein AJ, Moser KW, Thompson RC, Cerqueira MD, Henzlova MJ. Radiation dose to patients from cardiac diagnostic imaging. Circulation. 2007 Sep 11;116(11):1290-305. doi: 10.1161/CIRCULATIONAHA.107.688101. No abstract available. PMID 17846343
- [Result] Rochitte CE, George RT, Chen MY, Arbab-Zadeh A, Dewey M, Miller JM, Niinuma H, Yoshioka K, Kitagawa K, Nakamori S, Laham R, Vavere AL, Cerci RJ, Mehra VC, Nomura C, Kofoed KF, Jinzaki M, Kuribayashi S, de Roos A, Laule M, Tan SY, Hoe J, Paul N, Rybicki FJ, Brinker JA, Arai AE, Cox C, Clouse ME, Di Carli MF, Lima JA. Computed tomography angiography and perfusion to assess coronary artery stenosis causing perfusion defects by single photon emission computed tomography: the CORE320 study. Eur Heart J. 2014 May;35(17):1120-30. doi: 10.1093/eurheartj/eht488. Epub 2013 Nov 19. PMID 24255127